CLINICAL TRIAL: NCT04196816
Title: Surgery/Destruction for Stage IV Pancreatic Cancer With Oligo-Metastatic Disease
Brief Title: Surgery for Pancreatic Cancer With Oligo-Metastasis
Acronym: SPaM
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); Association de Chirurgie hepato-bilio-pancreatique et transplantation (ACHBT) (Unknown); Federation de recherche en chirurgie digestive (FRENCH) (Unknown); Club Français du Pancreas (CFP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0534
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer; Pancreatic Surgery
Keywords: Surgery; Metastasis surgery; Survival; Multimodal treatment; Stage IV
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic cancer is increasing in incidence and will be the second leading cause of cancer-related deaths in 2030 in the West. Only 10 to 15% of patients are eligible for curative resection with long-term survival rarely exceeding 20% at 5 years. The management of metastatic or recurrent diseases can not, unfortunately, be recommended to date because of limited data available (INCA 2019).

However, recent, low-strength publications have reported encouraging results on the long-term survival of stage IV or recurrent patients.

The aim of the present retrospective cohort study is to analyze results of surgery/destruction of metastatic synchronous or metachronous disease or local recurrence in patients with stage IV pancreatic cancer

ELIGIBILITY:
Inclusion criteria:

- Patients who had resection or destruction of one or more synchronous or metachronous metastases or local recurrence of pancreatic adenocarcinoma

Details:

* synchronous lesions, metachrones can be included
* all distant lesions (hepatic, pulmonary) can be included
* documented lymph node involvement after analysis of the specimen (hepatic hilum, mesenteric root, retroperitoneal or inter-aortic-cellar) can be included
* patients with local recurrence who underwent surgical treatment

Exclusion Criteria:

- Patient who reject the study protocol

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had resection or destruction of one or more synchronous or metachronous metastases or local recurrence of pancreatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival at 3 years (percentage of patients alive). Overall survival (OS) (time from diagnosis until death, regardless of cause)

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival (percentage of patients without recurrence) at 3 years. Progression-free survival (PFS) (time from diagnosis to time of first radiological evidence of local, regional, or distant relapse, or death due to any cause)

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC